CLINICAL TRIAL: NCT04004494
Title: Three-dimensional Computed Tomography Reconstruction for Operative Planning in VATS Segmentectomy
Brief Title: 3D Reconstruction in Video-assisted Thoracoscopic Surgery (VATS) Segmentectomy
Acronym: DRIVATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Union hospital of Fujian Medical University (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTS-008
Record Dates: First submitted 2019-06-23; First posted 2019-07-02 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Segmentectomy
Keywords: segmentectomy; Video-assisted thoracoscopic surgery; lung cancer; ground-glass opacity
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Reconstruction (Experimental): Chest contrast-enhanced computed tomography will be performed preoperatively, and 3-dimensional reconstruction will be formed based on the data of chest CT. Video-assisted segmentectomy will be performed guided by the image of 3-dimensional CT. IPS-lung software (Shenzhen Yorktal Digital Medical Imaging Technology Company, Shenzhen, China) will be used preoperatively to construct a 3D-image to ascertain the position and structure of targeted segmental blood vessels and bronchi.
  Interventions: Other: 3D reconstruction
- Chest computed tomography (No Intervention): Chest contrast-enhanced computed tomography will be performed preoperatively. Video-assisted segmentectomy will be performed based on the image of preoperative chest CT

INTERVENTIONS:
Other: 3D reconstruction — 3-dimensional computed tomography reconstruction guided VATS segmentectomy
  Arms: 3D Reconstruction

SUMMARY:
Anatomical variations of pulmonary vessel may cause serious problems during pulmonary segmentectomy. Three-dimensional （3D）computed tomography (CT) presents 3D images of pulmonary vessels and the tracheobronchial tree and may help operative planning. Retrospective studies have identified the importance of 3-dimensional CT in the field of pulmonary segmentectomy. And the aim of this study is to compare the usefulness of 3-dimensional CT with standard chest CT in preoperative planning of video-assisted segmentectomy.

DETAILED DESCRIPTION:
Lung cancer has been the most serious malignancy around the world which has the highest morbidity and mortality amount all the malignant tumors. Due to the wide spread of lung cancer screening, more and more early stage lung cancer patients have been diagnosed. Video-assisted segmentectomy is a standard surgical procedure in treating early stage peripheral non-small cell lung cancer (NSCLC). However, anatomical variations of pulmonary vessel may cause serious problems, for example unexpected bleed during surgery. Three-dimensional computed tomography (CT), which is reconstructed based on the standard chest CT image, presents 3D images of pulmonary vessels and the tracheobronchial tree and therefore helps operative planning. There are several retrospective studies addressed the importance of 3-dimensional CT in the field of pulmonary segmentectomy. And the aim of this multicenter randomized controlled trial is to compare the usefulness of 3-dimensional CT and standard chest CT in preoperative planning of video-assisted segmentectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 18 years;
2. Pulmonary nodules or ground glass opacification （GGO） found in chest CT examination, and conform with indications for segmentectomy:

   Peripheral nodule 0.8-2 cm with at least one of the following:

   i. Histology of adenocarcinoma in situ; ii. Nodule has ≥50% ground-glass appearance on CT; iii. Radiologic surveillance confirms a long doubling time (≥400 days). Segmentectomy should achieve parenchymal resection margins ≥2 cm or ≥ the size of the nodule.
3. Adequate cardiac function, respiratory function, liver function and renal function for anesthesia and VATS segmentectomy.
4. American Society of Anesthesiologists (ASA) score: Grade I-III.
5. Patients who can coordinate the treatment and research and sign the informed consent.

Exclusion Criteria:

1. Patients with a significant medical condition which is thought unlikely to tolerate the surgery. For example, cardiac disease, significant liver and renal function disorder.
2. Patients with psychiatric disease who are expected lack of compliance with the protocol.
3. Patients have history of chest trauma or surgery on ipsilateral chest which may cause pleural adhesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
operative time | During surgery
  the time of operation

SECONDARY OUTCOMES:
blood loss | During surgery
  Amount of intraoperative blood loss
conversion rate | During surgery
  the rate of conversion to open surgery in the operation
operative accident event | During surgery
  the accident event happened in operative. For example, a segmentectomy is converted to a lobectomy
Incidence of postoperative complications | Postoperative in-hospital stay up to 30 days
  mainly include: pneumonia, arrhythmia, incision infection, vocal cord paralysis, trachea cannula
Postoperative hospital stay | Up to 24 weeks
  length of stay in hospitalization
Duration of chest tube placement | Up to 4 weeks
  Duration of chest tube placement
30-day mortality | Postoperative in-hospital stay up to 30 days
  30-day mortality after surgery
dissection of lymph nodes | 2 weeks after surgery
  including overall lymph node count, number of stations dissected and number of lymph nodes in each lymph node station
Overall survival (OS) | up to 60 months
  Up to the date of death of any causes since the date of randomization
Disease-free survival （DFS） | up to 60 months
  Up to the date of disease recurrence since the date of randomization
Preoperative lung function | Baseline
  forced expiratory volume at one second（FEV1） in litre, maximal voluntary ventilation （MVV） in litre
Postoperative lung function | at the 3rd month after surgery
  forced expiratory volume at one second（FEV1） in litre, maximal voluntary ventilation （MVV） in litre
Incidence of change of surgical plan | During surgery
  Surgical plan is made based of the image of standard chest computed tomography or three-dimensional computed tomography, the targeted segmental bronchus and pulmonary vessels are decided preoperatively. Change of surgical plan is recorded when the actually resected bronchus and vessels are different to those in the preoperative surgical plan

OTHER OUTCOMES:
Total hospitalization expenditures | postoperative in-hospital stay up to 30 days
  cost in hospital
Anatomical variations | During surgery
  Rate of anatomical variation of segmental bronchus and pulmonary vessel in Chinese population

CONTACTS AND LOCATIONS:
Overall Officials: He-Cheng Li, doctor, Study Director — Ruijin Hospital
Locations (3):
- China (3):
  - Union Hospital of Fujian medical university, Fujian, Fujian
  - Guangdong General Hospital, Guangdong, Guangdong
  - Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niu Z, Chen K, Jin R, Zheng B, Gong X, Nie Q, Jiang B, Zhong W, Chen C, Li H. Three-dimensional computed tomography reconstruction in video-assisted thoracoscopic segmentectomy (DRIVATS): A prospective, multicenter randomized controlled trial. Front Surg. 2022 Oct 13;9:941582. doi: 10.3389/fsurg.2022.941582. eCollection 2022. PMID 36311929